CLINICAL TRIAL: NCT05380947
Title: Relative Bioavailability of BI 1810631 as Two Different Oral Formulations Given as Single Doses and Investigation of the Effects of Food and Multiple-dose Rabeprazole on the Pharmacokinetics of Single-dose BI 1810631 Following Oral Administration in Healthy Male Subjects (an Open-label, Randomised, Four-way Crossover Trial)
Brief Title: A Study in Healthy Men to Compare Two Different Oral Formulations of BI 1810631 and to Test How Food or Rabeprazole Influence the Amount of BI 1810631 in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1479-0003; 2022-000268-23 (EudraCT Number)
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Results first posted 2025-11-04 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Healthy
MeSH Terms: interventions — Rabeprazole

STUDY DESIGN:
Intervention Model Description: 4-way crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment sequence 1: R - T1 - T2 - T3 (Experimental): Treatments:
  R: TF1 fasted T1: NF fasted T2: NF fed T3: NF fasted + rabeprazole
  Interventions: Drug: BI 1810631 - trial formulation 1 (TF1); Drug: BI 1810631 - new formulation (NF); Drug: Rabeprazole sodium
- Treatment sequence 2: T1 - T3 - R - T2 (Experimental)
  Interventions: Drug: BI 1810631 - trial formulation 1 (TF1); Drug: BI 1810631 - new formulation (NF); Drug: Rabeprazole sodium
- Treatment sequence 3: T2 - R - T3 - T1 (Experimental)
  Interventions: Drug: BI 1810631 - trial formulation 1 (TF1); Drug: BI 1810631 - new formulation (NF); Drug: Rabeprazole sodium
- Treatment sequence 4: T3 - T2 - T1 - R (Experimental)
  Interventions: Drug: BI 1810631 - trial formulation 1 (TF1); Drug: BI 1810631 - new formulation (NF); Drug: Rabeprazole sodium

INTERVENTIONS:
Drug: BI 1810631 - trial formulation 1 (TF1) — BI 1810631 - trial formulation 1 (TF1)
  Other Names: Zongertinib,; Hernexeos®
Drug: BI 1810631 - new formulation (NF) — BI 1810631 - new formulation (NF)
  Other Names: Zongertinib,; Hernexeos®
Drug: Rabeprazole sodium — Rabeprazole sodium
  Other Names: Pariet®

SUMMARY:
BI 1810631 trial formulation 1 (TF1) is currently used in clinical trials, but is planned to be replaced by another formulation (principle) in future clinical trials and on the market. This trial intends to bridge pharmacokinetics (PK) between the two formulation principles. For this, relative bioavailability of TF1 and new formulation (NF) is assessed. Moreover the trial intends to inform on the effect of food and of the proton pump inhibitor rabeprazole on the PK of BI 1810631 after administration as NF in order to inform management of food and concomitant medications.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (Blood pressure (BP), Pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 45 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 weight divided by height squared (kg/m2) (inclusive)
* Signed and dated written informed consent in accordance with International Council on Harmonisation - Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial

Exclusion Criteria:

* Any finding in the medical examination (including blood pressure (BP), pulse rate (PR) or electrocardiogram (ECG)) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetre of mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* further exclusion criteria apply

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2022-06-23 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization). For more details refer to: https:// www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was to investigate the relative bioavailability of 2 different BI 1810631 oral formulations (trial formulation 1 [TF1], Reference [R] and new formulation [NF], Test 1 [T1]) under fasting conditions; BI 1810631 NF under fasting (T1) and fed (T2) conditions; BI 1810631 NF given alone (T1) and together with the proton pump inhibitor rabeprazole (T3) under fasting conditions.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria.
  Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Treatment Sequence 1: R - T1 - T2 - T3: The treatment sequence R-T1-T2-T3 was administered. The treatments were separated by a washout interval of at least 14 days between BI 1810631 administrations.
  Reference (R): 30 mg BI 1810631 as trial formulation 1 (TF1) were administered orally as single dose once on Day 1 of respective period under fasted condition.
  Test 1 (T1): 30 mg BI 1810631 as new formulation (NF) were administered orally as single dose once on Day 1 of respective period under fasted condition.
  T2: 30 mg BI 1810631 as NF were administered orally as single dose once on Day 1 of respective period under fed condition.
  T3: 2 gastroresistant tablets of 20 mg Pariet® (rabeprazole; 40 mg per dose) were administered orally once daily over Day -4 to Day 1 (5 days in total) of respective period; 30 mg BI 1810631 as NF were administered orally as single dose once on Day 1 of respective period under fasted condition.
- Treatment Sequence 2: T1 - T3 - R - T2: The treatment sequence T1 - T3 - R - T2 was administered. The treatments were separated by a washout interval of at least 14 days between BI 1810631 administrations.
  Reference (R): 30 mg BI 1810631 as trial formulation 1 (TF1) were administered orally as single dose once on Day 1 of respective period under fasted condition.
  Test 1 (T1): 30 mg BI 1810631 as new formulation (NF) were administered orally as single dose once on Day 1 of respective period under fasted condition.
  T2: 30 mg BI 1810631 as NF were administered orally as single dose once on Day 1 of respective period under fed condition.
  T3: 2 gastroresistant tablets of 20 mg Pariet® (rabeprazole; 40 mg per dose) were administered orally once daily over Day -4 to Day 1 (5 days in total) of respective period; 30 mg BI 1810631 as NF were administered orally as single dose once on Day 1 of respective period under fasted condition.
- Treatment Sequence 3: T2 - R - T3 - T1: The treatment sequence T2 - R - T3 - T1 was administered. The treatments were separated by a washout interval of at least 14 days between BI 1810631 administrations.
  Reference (R): 30 mg BI 1810631 as trial formulation 1 (TF1) were administered orally as single dose once on Day 1 of respective period under fasted condition.
  Test 1 (T1): 30 mg BI 1810631 as new formulation (NF) were administered orally as single dose once on Day 1 of respective period under fasted condition.
  T2: 30 mg BI 1810631 as NF were administered orally as single dose once on Day 1 of respective period under fed condition.
  T3: 2 gastroresistant tablets of 20 mg Pariet® (rabeprazole; 40 mg per dose) were administered orally once daily over Day -4 to Day 1 (5 days in total) of respective period; 30 mg BI 1810631 as NF were administered orally as single dose once on Day 1 of respective period under fasted condition.
- Treatment Sequence 4: T3 - T2 - T1 - R: The treatment sequence T3 - T2 - T1 - R was administered. The treatments were separated by a washout interval of at least 14 days between BI 1810631 administrations.
  Reference (R): 30 mg BI 1810631 as trial formulation 1 (TF1) were administered orally as single dose once on Day 1 of respective period under fasted condition.
  Test 1 (T1): 30 mg BI 1810631 as new formulation (NF) were administered orally as single dose once on Day 1 of respective period under fasted condition.
  T2: 30 mg BI 1810631 as NF were administered orally as single dose once on Day 1 of respective period under fed condition.
  T3: 2 gastroresistant tablets of 20 mg Pariet® (rabeprazole; 40 mg per dose) were administered orally once daily over Day -4 to Day 1 (5 days in total) of respective period; 30 mg BI 1810631 as NF were administered orally as single dose once on Day 1 of respective period under fasted condition.
Period: Period 1
Arm/Group | Treatment Sequence 1: R - T1 - T2 - T3 | Treatment Sequence 2: T1 - T3 - R - T2 | Treatment Sequence 3: T2 - R - T3 - T1 | Treatment Sequence 4: T3 - T2 - T1 - R
Started | 3 | 4 | 3 | 3
Completed | 3 | 4 | 3 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period 1
Arm/Group | Treatment Sequence 1: R - T1 - T2 - T3 | Treatment Sequence 2: T1 - T3 - R - T2 | Treatment Sequence 3: T2 - R - T3 - T1 | Treatment Sequence 4: T3 - T2 - T1 - R
Started | 3 | 4 | 3 | 3
Completed | 2 | 4 | 3 | 3
Not Completed | 1 | 0 | 0 | 0
Not completed — Not attend visit | 1 | 0 | 0 | 0
Period: Period 2
Arm/Group | Treatment Sequence 1: R - T1 - T2 - T3 | Treatment Sequence 2: T1 - T3 - R - T2 | Treatment Sequence 3: T2 - R - T3 - T1 | Treatment Sequence 4: T3 - T2 - T1 - R
Started | 2 | 4 | 3 | 3
Completed | 2 | 4 | 3 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period 2
Arm/Group | Treatment Sequence 1: R - T1 - T2 - T3 | Treatment Sequence 2: T1 - T3 - R - T2 | Treatment Sequence 3: T2 - R - T3 - T1 | Treatment Sequence 4: T3 - T2 - T1 - R
Started | 2 | 4 | 3 | 3
Completed | 1 | 4 | 3 | 3
Not Completed | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Period: Period 3
Arm/Group | Treatment Sequence 1: R - T1 - T2 - T3 | Treatment Sequence 2: T1 - T3 - R - T2 | Treatment Sequence 3: T2 - R - T3 - T1 | Treatment Sequence 4: T3 - T2 - T1 - R
Started | 1 | 4 | 3 | 3
Completed | 1 | 4 | 3 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period 3
Arm/Group | Treatment Sequence 1: R - T1 - T2 - T3 | Treatment Sequence 2: T1 - T3 - R - T2 | Treatment Sequence 3: T2 - R - T3 - T1 | Treatment Sequence 4: T3 - T2 - T1 - R
Started | 1 | 4 | 3 | 3
Completed | 1 | 2 | 3 | 2
Not Completed | 0 | 2 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Not attend visit | 0 | 1 | 0 | 1
Period: Period 4
Arm/Group | Treatment Sequence 1: R - T1 - T2 - T3 | Treatment Sequence 2: T1 - T3 - R - T2 | Treatment Sequence 3: T2 - R - T3 - T1 | Treatment Sequence 4: T3 - T2 - T1 - R
Started | 1 | 2 | 3 | 2
Completed | 1 | 2 | 3 | 2
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): the TS included all subjects who were treated with at least one dose of trial drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence 1: R - T1 - T2 - T3 | Treatment Sequence 2: T1 - T3 - R - T2 | Treatment Sequence 3: T2 - R - T3 - T1 | Treatment Sequence 4: T3 - T2 - T1 - R | Total
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 13
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.7 (7.0) | 33.5 (3.1) | 34.7 (8.5) | 34.0 (7.2) | 34.8 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 3 | 4 | 3 | 3 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 4 | 3 | 3 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 1
  White | 3 | 3 | 3 | 3 | 12
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of BI 1810631 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: The area under the concentration-time curve of BI 1810631 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) was reported.
  Unit of geometric coefficient of variation (gCV) is %.
Time Frame: Within 3 hours prior and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 34, 46, 70, 94 and 118 hours after BI 1810631 administration.
Population: Pharmacokinetic (PK) parameter analysis set (PKS): this set included all subjects in the treated set who provided at least 1 PK endpoint that was defined as primary or secondary and was not excluded due to a protocol violation relevant to the evaluation of PK or due to PK non-evaluability. Only participants with non-missing results were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour * nanomole / Liter (h*nmol/L)
Groups:
- TF1 Fasted (R): Reference (R): 30 mg BI 1810631 as trial formulation 1 (TF1) were administered orally as single dose once on Day 1 of respective period under fasted condition.
- NF Fasted (T1): Test 1 (T1): 30 mg BI 1810631 as new formulation (NF) were administered orally as single dose once on Day 1 of respective period under fasted condition.
- NF Fed (T2): Test 2 (T2): 30 mg BI 1810631 as new formulation (NF) were administered orally as single dose once on Day 1 of respective period under fed condition.
- NF Fasted + Rabeprazole (T3): Test 3 (T3): 2 gastroresistant tablets of 20 milligrams (mg) Pariet® (rabeprazole; 40 mg per dose) were administered orally once daily over Day -4 to Day 1 (5 days in total) of respective period; 30 mg BI 1810631 as new formulation (NF) were administered orally as single dose once on Day 1 of respective period under fasted condition.
Arm/Group | TF1 Fasted (R) | NF Fasted (T1) | NF Fed (T2) | NF Fasted + Rabeprazole (T3)
Number analyzed (Participants) | 12 | 12 | 9 | 11
hour * nanomole / Liter (h*nmol/L) | 4240 (52.7) | 5680 (18.8) | 4060 (13.7) | 5410 (27.6)
Statistical Analysis 1: Comparison: TF1 Fasted (R) vs NF Fasted (T1); Test type: Other — The statistical model was an analysis of variance (ANOVA) model on the logarithmic scale including effects for sequence, subjects nested within sequences, period, and treatment. The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed; Adjusted geometric means ratio (T1/R) = 135.2, 90% CI 2-sided [99.7 to 183.6] — Unit of adjusted geometric means ratio (T1/R) is %. Unit of 90% Confidence Interval is %. Intra-individual geometric coefficient of variation (gCV) = 39.7%
Statistical Analysis 2: Comparison: NF Fasted (T1) vs NF Fed (T2); Test type: Other — [test comment as in outcome 1, analysis 1]; Adjusted geometric means ratio (T2/T1) = 74.2, 90% CI 2-sided [67.6 to 81.6] — Unit of adjusted geometric means ratio (T2/T1) is %. Unit of 90% Confidence Interval is %. Intra-individual geometric coefficient of variation (gCV) = 9.8%
Statistical Analysis 3: Comparison: NF Fasted (T1) vs NF Fasted + Rabeprazole (T3); Test type: Other — [test comment as in outcome 1, analysis 1]; Adjusted geometric means ratio (T3/T1) = 97.1, 90% CI 2-sided [85.8 to 110.0] — Unit of adjusted geometric means ratio (T3/T1) is %. Unit of 90% Confidence Interval is %. Intra-individual geometric coefficient of variation (gCV) = 13.8%

2. Primary Outcome: Maximum Measured Concentration of BI 1810631 in Plasma (Cmax)
Description: The maximum measured concentration of BI 1810631 in plasma (Cmax) was reported.
  Unit of geometric coefficient of variation (gCV) is %.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole / Liter (nmol/L)
Arm/Group | TF1 Fasted (R) | NF Fasted (T1) | NF Fed (T2) | NF Fasted + Rabeprazole (T3)
Number analyzed (Participants) | 12 | 12 | 9 | 11
nanomole / Liter (nmol/L) | 291 (93.1) | 399 (37.3) | 208 (31.4) | 327 (34.2)
Statistical Analysis 1: Comparison: TF1 Fasted (R) vs NF Fasted (T1); Test type: Other — [test comment as in outcome 1, analysis 1]; Adjusted geometric means ratio (T1/R) = 139.3, 90% CI 2-sided [87.7 to 221.3] — Unit of adjusted geometric means ratio (T1/R) is %. Unit of 90% Confidence Interval is %. Intra-individual coefficient of variation (gCV) = 62.3%
Statistical Analysis 2: Comparison: NF Fasted (T1) vs NF Fed (T2); Test type: Other — [test comment as in outcome 1, analysis 1]; Adjusted geometric means ratio (T2/T1) = 53.5, 90% CI 2-sided [40.5 to 70.8] — Unit of adjusted geometric means ratio (T2/T1) is %. Unit of 90% Confidence Interval is %. Intra-individual coefficient of variation (gCV) = 31.0%
Statistical Analysis 3: Comparison: NF Fasted (T1) vs NF Fasted + Rabeprazole (T3); Test type: Other — [test comment as in outcome 1, analysis 1]; Adjusted geometric means ratio (T3/T1) = 87.0, 90% CI 2-sided [66.8 to 113.2] — Unit of adjusted geometric means ratio (T3/T1) is %. Unit of 90% Confidence Interval is %. Intra-individual coefficient of variation (gCV) = 30.5%

3. Secondary Outcome: Area Under the Concentration-time Curve of BI 1810631 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: The area under the concentration-time curve of BI 1810631 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) was reported.
  Unit of geometric coefficient of variation (gCV) is %.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour * nanomole / Liter (h * nmol/L)
Arm/Group | TF1 Fasted (R) | NF Fasted (T1) | NF Fed (T2) | NF Fasted + Rabeprazole (T3)
Number analyzed (Participants) | 11 | 12 | 9 | 11
hour * nanomole / Liter (h * nmol/L) | 4550 (52.7) | 5980 (19.2) | 4310 (14.2) | 5660 (28.8)
Statistical Analysis 1: Comparison: TF1 Fasted (R) vs NF Fasted (T1); Test type: Other — [test comment as in outcome 1, analysis 1]; Adjusted geometric means ratio (T1/R) = 129.1, 90% CI 2-sided [96.2 to 173.4] — Unit of adjusted geometric means ratio (T1/R) is %. Unit of 90% Confidence Interval is %. Intra-individual coefficient of variation (gCV) =36.6%
Statistical Analysis 2: Comparison: NF Fasted (T1) vs NF Fed (T2); Test type: Other — [test comment as in outcome 1, analysis 1]; Adjusted geometric means ratio (T2/T1) = 74.9, 90% CI 2-sided [68.6 to 81.7] — Unit of adjusted geometric means ratio (T2/T1) is %. Unit of 90% Confidence Interval is %. Intra-individual coefficient of variation (gCV) = 9.0%
Statistical Analysis 3: Comparison: NF Fasted (T1) vs NF Fasted + Rabeprazole (T3); Test type: Other — [test comment as in outcome 1, analysis 1]; Adjusted geometric means ratio (T3/T1) = 96.9, 90% CI 2-sided [85.3 to 110.2] — Unit of adjusted geometric means ratio (T3/T1) is %. Unit of 90% Confidence Interval is %. Intra-individual coefficient of variation (gCV) = 14.2%

ADVERSE EVENTS:
Time Frame: For R, T1, T2, and NF fasted + Rabeprazole (Rab.): From drug administration (admin.) till end of 14-day residual effect period (REP), up to 14 days. For Rab.: From drug admin. till end of REP of Rab., up to 8 days. All-cause mortality: From the first drug administration till end of trial, up to a total of 64 days.
Description: Treated set (TS): the TS included all subjects who were treated with at least one dose of trial drug.
Groups:
- Rabeprazole: 2 gastroresistant tablets of 20 milligrams (mg) Pariet® (rabeprazole; 40 mg per dose) were administered orally once daily over Day -4 to Day 1 (5 days in total) of respective period.
Arm/Group | TF1 Fasted (R) | NF Fasted (T1) | NF Fed (T2) | Rabeprazole | NF Fasted + Rabeprazole (T3)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/9 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/9 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 4/12 | 1/12 | 4/9 | 2/11 | 4/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TF1 Fasted (R) (N=12) | NF Fasted (T1) (N=12) | NF Fed (T2) (N=9) | Rabeprazole (N=11) | NF Fasted + Rabeprazole (T3) (N=11)
COVID-19 (Infections and infestations) | 2 | 1 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-05-25): https://cdn.clinicaltrials.gov/large-docs/47/NCT05380947/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-17): https://cdn.clinicaltrials.gov/large-docs/47/NCT05380947/SAP_001.pdf